CLINICAL TRIAL: NCT00408109
Title: VRC 304: A Phase I Study of the Safety and Immunogenicity of a Recombinant DNA Plasmid Vaccine (VRC-AVIDNA036-00-VP), Encoding for the Influenza Virus H5 Hemagglutinin Protein in Healthy Adults
Brief Title: Safety Study of Avian Flu Vaccine
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 070042; 07-I-0042
Record Dates: First submitted 2006-12-05; First posted 2006-12-06 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2008-08-28

CONDITIONS: Influenza A Virus, H5N1 Subtype; Influenza A Virus; Influenzavirus A; Orthomyxoviridae; H5N1 Virus
Keywords: Avian Influenza; Healthy; Immunity; Preventive; Bird Flu; Healthy Volunteer; HV
MeSH Terms: conditions — Influenza in Birds

INTERVENTIONS:
Drug: VRC-AVIDNA036-00-VP

SUMMARY:
This study will determine if an experimental avian flu (bird flu) vaccine is safe, whether it has side effects and if it can stimulate an immune response in people. The vaccine being tested in this study is made from DNA (genetic material) that codes for an influenza protein called hemagglutinin 5 (H5), which is based on the protein from the bird flu virus. The study will determine if the body creates resistance or immunity to the H5 protein. The hope is that an immune response to this protein may protect against bird flu virus infection.

Healthy people between 18 and 60 years old who have been vaccinated with the current season's influenza vaccine may be eligible for this study.

Participants are randomly assigned to receive injections of one of the following: 1) study vaccine at 1 mg dose, 2) study vaccine at 4 mg dose, or 3) placebo (salt-water solution). They receive three injections about 4 weeks apart in the upper arm muscle. Participants record their temperature and symptoms at home for 5 days after each injection, either on a diary card or electronically using the Internet, and report any side effects to a study physician or nurse as soon as possible. They return to NIH for clinic visits every 2 weeks for the first 12 weeks, then at week 26 and at week 42 to check for health changes or problems. Blood is drawn at all visits and urine samples are collected through week 10.

If a participant develops serious side effects, the study physician may decide that he or she should not receive any further injections. However, all participants are asked to continue the follow-up visits even if they do not get the full set of three injections.

...

DETAILED DESCRIPTION:
Study Design: This is a Phase I double-blind, placebo-controlled study to evaluate safety, tolerability, and immunogenicity of a recombinant DNA vaccine against the influenza virus hemagglutinin H5. The hypothesis is that this vaccine will be safe for human administration and will elicit antibody and T cell responses against the H5 protein. The primary objectives are to evaluate the safety and tolerability of the investigational vaccine at a 1-mg and 4-mg dose in healthy adults. Secondary and exploratory objectives are related to the immunogenicity of the study vaccine.

Product Description: The vaccine is composed of a single closed-circular DNA plasmid that encodes the H5 protein with a CMV/R promoter. Vaccine vials will be supplied at 4 mg/mL. Each vaccination will be 1 mL administered intramuscularly (IM) in the deltoid muscle using the Biojector 2000 Needle-Free Injection Management System (Biojector). The placebo and diluent is phosphate buffered saline (PBS).

Subjects: A total of 45 healthy adults, ages 18-60 years, will be enrolled.

Study Plan: Subjects will be simultaneously randomized at a ratio of 1:1:1 into one of two dosage groups or a placebo group. Subjects and clinicians will be blinded to group assignment. All subjects will receive 3 injections on the schedule shown in the schema. The protocol requires nine clinic visits and three telephone follow-up contacts.

Study Duration: Each participant will complete 42 weeks of clinical follow up.

Study Endpoints: The primary endpoint is safety and tolerability of the regimen. The secondary immunogenicity endpoint is H5-specific antibody as measured by hemagglutination inhibition (HAI) assay at Study Week 12. H5-specific T cell responses measured by intracellular cytokine staining (ICS) assay, enzyme-linked immunospot (ELISPOT) assays and other immunogenicity assays at timepoints throughout the study may also be completed as exploratory evaluations.

ELIGIBILITY:
* INCLUSION CRITERIA:

A participant must meet all of the following criteria:

1. 18 to 60 years old.
2. Available for clinical follow-up through Week 42.
3. Immunized with the current season FDA-approved influenza vaccine prior to enrollment at the specified interval [14 days to 24 weeks prior to enrollment for the inactivated influenza vaccine OR 30 days to 24 weeks prior to enrollment for the live-attenuated influenza vaccine (FluMist)].
4. Able to provide proof of identity to the satisfaction of the study clinician completing the enrollment process.
5. Complete an AoU prior to enrollment and verbalize understanding of all questions answered incorrectly.
6. Able and willing to complete the informed consent process.
7. Willing to donate blood for sample storage to be used for future research.
8. In good general health without clinically significant medical history.
9. Physical examination and laboratory results without clinically significant findings and a Body Mass Index (BMI) less than 40 within the 28 days prior to enrollment.

   Laboratory Criteria within 28 days prior to enrollment:
10. Hemoglobin greater than or equal to 11.5 g/dL for women; greater than or equal to 13.5 g/dL for men.
11. White blood cells (WBC) equal 3,300-12,000 cells/mm(3).
12. Differential either within institutional normal range or accompanied by site physician approval.
13. Total lymphocyte count greater than or equal to 800 cells/mm(3).
14. Platelets equal 125,000 - 400,000/mm(3).
15. Alanine aminotransferase (ALT) less than or equal to 1.25 times the upper limit of normal.
16. Serum creatinine less than or equal to 1 x upper limits of normal (less than or equal to 1.3 mg/dL for females; less than or equal to 1.4 mg/dL for males).
17. Normal urinalysis, defined as negative glucose, negative or trace protein and no clinically significant blood in the urine.
18. Negative FDA-approved HIV blood test. [Note: Results of HIV enzyme-linked immunosorbent assay (ELISA) will be documented, but a negative HIV polymerase chain reaction (PCR) test result will be sufficient for eligibility screening of subjects with positive HIV ELISA that is due to prior participation in an HIV vaccine study].
19. Negative hepatitis B surface antigen (HBsAg)
20. Negative anti-hepatitis C virus (HCV) antibody and negative HCV PCR.

    Female-Specific Criteria:
21. Negative beta-HCG pregnancy test (urine or serum) for women presumed to be of reproductive potential.
22. A female participant must meet one of the following criteria:

No reproductive potential because of menopause [one year without menses] or because of a hysterectomy, bilateral oophorectomy, or tubal ligation,

OR

Participant agrees to be heterosexually inactive at least 21 days prior to enrollment and through Week 26 of the study,

OR

Participant agrees to consistently practice contraception at least 21 days prior to enrollment and through Week 26 of the study by one of the following methods: condoms, male or female, with or without a spermicide; diaphragm or cervical cap with spermicide; intrauterine device; contraceptive pills, patch, implant or any other FDA-approved contraceptive method; male partner has previously undergone a vasectomy.

EXCLUSION CRITERIA:

A volunteer will be excluded if one or more of the following conditions apply.

Women Specific:

1. Breast-feeding or planning to become pregnant during the study.

   Volunteer has received any of the following substances:
2. Immunosuppressive medications, cytotoxic medications, inhaled corticosteroids, or long-acting beta-agonists within the past three months. [With the exceptions that use of corticosteroid nasal spray for rhinitis; topical corticosteroids for an acute uncomplicated dermatitis; short-acting beta-agonist use in controlled asthmatics; or a short course (10 days or less) of corticosteroids for a non-chronic condition at least 2 weeks prior to enrollment in this study will not exclude study participation.]
3. Blood products within 120 days prior to HIV screening.
4. Immunoglobulin within 60 days prior to HIV screening.
5. Live attenuated vaccines within 30 days prior to initial study vaccine administration.
6. Investigational research agents within 30 days prior to initial study vaccine administration.
7. Medically indicated subunit or killed vaccines, e.g. influenza, pneumococcal, or allergy treatment with antigen injections, within 14 days of study vaccine administration.
8. Current anti-TB prophylaxis or therapy.
9. Previous H5 avian influenza investigational vaccine.

   Volunteer has a history of any of the following clinically significant conditions:
10. Autoimmune disease or immunodeficiency.
11. Contraindication to receiving an FDA approved 2006-2007 seasonal influenza vaccination (e.g., egg allergy).
12. Serious adverse reactions to vaccines such as anaphylaxis, urticaria (hives), respiratory difficulty, angioedema, or abdominal pain.
13. A history of hereditary angioedema (HAE), acquired angioedema (AAE), or idiopathic forms of angioedema.
14. Asthma that is unstable or required emergent care, urgent care, hospitalization or intubation during the past two years or that requires the use of oral or intravenous corticosteroids.
15. Diabetes mellitus (type I or II), with the exception of gestational diabetes.
16. History of thyroidectomy or thyroid disease that required medication within the past 12 months.
17. Idiopathic urticaria within the past 2 years.
18. Hypertension that is not well controlled by medication or is more than 145/95 at enrollment.
19. Bleeding disorder diagnosed by a doctor (e.g. factor deficiency, coagulopathy, or platelet disorder requiring special precautions) or significant bruising or bleeding difficulties with IM injections or blood draws.
20. Malignancy that is active or treated malignancy for which there is not reasonable assurance of sustained cure or malignancy that is likely to recur during the period of the study.
21. Seizure disorder other than: 1) febrile seizures under the age of two, 2) seizures secondary to alcohol withdrawal more than 3 years ago, or 3) a singular seizure not requiring treatment within the last 3 years.
22. Asplenia, functional asplenia or any condition resulting in the absence or removal of the spleen.
23. Allergic reaction to aminoglycoside antibiotics.
24. Psychiatric condition that precludes compliance with the protocol; past or present psychoses; past or present bipolar disorder; disorder requiring lithium; or within five years prior to enrollment, a history of suicide plan or attempt.
25. Any medical, psychiatric, social condition, occupational reason or other responsibility that, in the judgment of the investigator, is a contraindication to protocol participation or impairs a volunteer's ability to give informed consent.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 45
Dates: Start 2006-12-04; Study Completion 2008-08-28

PRIMARY OUTCOMES:
Safety (local and systemic reactogenicity, lab tests, AEs)

SECONDARY OUTCOMES:
Immunogenicity (cellular and humoral immune function assays)

CONTACTS AND LOCATIONS:
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Subbarao K, Murphy BR, Fauci AS. Development of effective vaccines against pandemic influenza. Immunity. 2006 Jan;24(1):5-9. doi: 10.1016/j.immuni.2005.12.005. PMID 16413916
- [Background] Luke CJ, Subbarao K. Vaccines for pandemic influenza. Emerg Infect Dis. 2006 Jan;12(1):66-72. doi: 10.3201/eid1201.051147. PMID 16494720
- [Background] Taubenberger JK, Reid AH, Lourens RM, Wang R, Jin G, Fanning TG. Characterization of the 1918 influenza virus polymerase genes. Nature. 2005 Oct 6;437(7060):889-93. doi: 10.1038/nature04230. PMID 16208372